CLINICAL TRIAL: NCT07203092
Title: Effects of Transcranial Photobiomodulation on Cognition and Brain Metabolism in Adults With ADHD
Brief Title: Effects of Transcranial Photobiomodulation in ADHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Francisco Gonzalez-Lima, PhD, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00007909
Record Dates: First submitted 2025-09-15; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; transcranial photobiomodulation; cognition; prefrontal cortex; brain metabolism
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active transcranial photobiomodulation (Active Comparator): Participants in this arm will receive active transcranial photobiomodulation to the forehead, targeting prefrontal cortex.
  Interventions: Device: Active transcranial photobiomodulation
- Sham transcranial photobiomodulation (Sham Comparator): Participants in this arm will undergo this same procedure as the active group, but with no 1064-nm light emitted by the device.
  Interventions: Device: Sham transcranial photobiomodulation

INTERVENTIONS:
Device: Active transcranial photobiomodulation — Active transcranial photobiomodulation to the forehead targeting prefrontal cortex involves administration of 1064-nm light delivered via laser with a 4 centimeter beam diameter and 250 mW/cm2 power density for 8 minutes per treatment.
  Arms: Active transcranial photobiomodulation
Device: Sham transcranial photobiomodulation — Identical procedure as active group, but without 1064-nm light emitted by the device.
  Arms: Sham transcranial photobiomodulation

SUMMARY:
The investigators have previously shown that non-invasive methods of brain stimulation such as the administration of transcranial infrared light to the prefrontal cortex (PFC) can result in improvements to cognition and emotion as well as brain oxygenation. This method is called transcranial photobiomodulation (tPBM).

The investigators hypothesize that tPBM can improve cognition and brain oxygenation in adults with attention deficit hyperactivity disorder (ADHD). The investigators will investigate the effects of repeated tPBM sessions on cognitive functioning in adults with ADHD. Specifically, the investigators hypothesize that participants that receive tPBM will show improvements in response control, sustained attention, and working memory, as well as improvements in prefrontal hemodynamics and a reduction in ADHD symptoms.

DETAILED DESCRIPTION:
This will be a double-blind, sham-controlled study to evaluate the neurobehavioral and PFC neurometabolic effects of repeated tPBM sessions in adults with ADHD. Adults with a history of medically-diagnosed ADHD will be recruited. Participants will be randomized to two arms: (1) active tPBM or (2) sham tPBM. All participants will complete three in-person sessions and one remote follow-up visit conducted online. Participant will receive three weekly sessions of tPBM targeting the PFC using a 1064 nm laser. Cognitive performance will be assessed using the continuous performance task and 2-back task at baseline and after the final tPBM session. The investigators predict that participants receiving active tPBM will show improvements in sustained attention, impulse control, and working memory. Functional near-infrared spectroscopy recordings, collected at baseline and post-treatment, will be used to evaluate changes in PFC hemodynamic response and network interactions (functional connectivity). The investigators predict that active tPBM will enhance the PFC hemodynamic response and strengthen network interactions across prefrontal subregions. Lastly, ADHD symptomatology will be assessed using the Adult ADHD Self-Report Scale at baseline, post-treatment, and at a four-week follow-up after tPBM. The investigators predict that participants receiving active tPBM will report progressive reductions in ADHD symptoms across time points.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Adults of any sex
* Age range: 18-44 years
* Any ethnic/racial background
* Medical history of ADHD
* Participants may either be on a stable ADHD medication regimen (with no changes within two weeks prior to the study) or not taking medication.

Exclusion Criteria:

* Currently pregnancy
* Any sham or active photobiomodulation treatment within the past five weeks.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Performance on the Continuous Performance Task | 1. Pre-Treatment: Baseline (Visit 1). 2. Post-treatment: Two weeks later (Visit 3).
  The Continuous Performance Task is a widely-used cognitive measure to evaluate sustained attention, vigilance, and response control. Participants respond to letters presented on a computer screen and inhibit their responses to the letter X. There is no score on a scale. An increase in Correct Rejections on CPT = better inhibition = better outcome of treatment.
Prefrontal oxygenation (functional near-infrared spectroscopy) | 1. Pre-Treatment: Baseline (Visit 1). 2. Post-treatment: Two weeks later (Visit 3).
  Participants will wear a head-mounted functional near-infrared spectroscopy device that records changes in the concentrations of oxygenated hemoglobin potentially resulting from the treatment.
Scores on the Adult ADHD Self-Report Scale (ASRS) questionnaire | 1. Pre-Treatment: Baseline (Visit 1). 2. Post-treatment: Two weeks later (Visit 3). 3. Follow-up: Four weeks later (Online).
  The ASRS is an 18-question self-assessment tool created by the World Health Organization (WHO) which evaluates symptom severity of ADHD. Minimum score=18; maximum score=90; high score = more ADHD symptoms; lower score after treatment = better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
What data will be shared? Individual participant data that underlie the results reported in this study, after deidentification (text, tables, figures, and appendices).
  A data dictionary, including a description of the variables and types of data, collected for each individual, will be provided. This data will include anonymized individual participant demographic information and all outcome variables (cognitive task data, spectroscopy data).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The raw data will be made available by the researchers upon reasonable request by any qualified doctoral researcher (PhD, MD). They will be granted access by contacting the corresponding author/principal investigator (F. Gonzalez-Lima, utbrainproject@gmail.com).
  It will be made available to qualified researchers whose proposed use of the data has been approved by an independent review committee (Institutional Review Board) identified for the purpose of individual participant data meta-analysis.
  Proposals may be submitted up to 36 months following article publication. After 36 months, the data will be available in our University's shared network drive, but without investigator support other than deposited metadata.
URL: https://labs.la.utexas.edu/gonzalez-lima/idp-plan/